CLINICAL TRIAL: NCT01074905
Title: A Randomised Open Label Study Comparing the Efficacy of Chloroquine/Primaquine, Chloroquine and Artesunate in the Treatment of Vivax Malaria Along the Thai-Burmese Border
Brief Title: Study on the Treatment of Vivax Malaria
Acronym: VHX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMRU0908
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Vivax Malaria
Keywords: vivax malaria; artesunate; chloroquine; primaquine; relapse
MeSH Terms: conditions — Malaria, Vivax; Recurrence | interventions — Artesunate; Chloroquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artesunate (Active Comparator): 2 mg/kg/day as single daily dose given for 5 days; maximum dose range is 1.6 to 2.4 mg/kg/day or a total of 8 to 12 mg/kg.
  Interventions: Drug: Artesunate
- Chloroquine (Active Comparator): 25 mg base/kg given in divided doses (10,10,5) over 3 days; Absolute range 20-30 mg/kg.
  Interventions: Drug: Chloroquine
- Chloroquine/Primaquine (Experimental): Chloroquine 3 days and Primaquine 14 days
  Interventions: Drug: Chloroquine/Primaquine

INTERVENTIONS:
Drug: Artesunate — 2 mg/kg/day as single daily dose given for 5 days; maximum dose range is 1.6 to 2.4 mg/kg/day or a total of 8 to 12 mg/kg.
  Arms: Artesunate
Drug: Chloroquine — 25 mg base/kg given in divided doses (10,10,5) over 3 days; Absolute range 20-30 mg/kg.
  Arms: Chloroquine
Drug: Chloroquine/Primaquine — Chloroquine 3 days and Primaquine 14 days
  Arms: Chloroquine/Primaquine

SUMMARY:
This is a randomised open label trial with follow up for 1 year. 660 adults and children above 6 months diagnosed with acute Plasmodium vivax will be randomised into 3 groups, either chloroquine, artesunate, or chloroquine/primaquine therapy. Participants will be screened on the day of inclusion then followed weekly for 8 visits and every 4 weeks until week 52. The primary objective of the study is to compare the efficacy of the WHO and Thai Ministry of Public Health recommended radical curative regimen of chloroquine and primaquine with the currently used monotherapy regimens of chloroquine and artesunate along the Thai-Burmese border.

DETAILED DESCRIPTION:
Considerably less attention has been paid to Plasmodium vivax epidemiology than Plasmodium falciparum. In areas of relatively low unstable transmission, which comprise the majority of P.vivax affected areas, vivax malaria is predominantly a disease of children (Luxemburger et al 1999). Chloroquine has long been the standard treatment for vivax malaria. Primaquine is recommended for radical cure of vivax malaria, but is difficult to administer due to dosing duration and side effects.

This study aims to characterize the epidemiologic history comparing the efficacy of 3 antimalarial regimens (chloroquine, artesunate, and chloroquine/primaquine) for plasmodium vivax in western Thailand. Chloroquine is currently the standard of treatment for Plasmodium vivax. Due to the long half-life or chloroquine, the first relapse of vivax malaria may be delayed. In contrast, artesunate has a very short half-life, thus, having no impact on first relapse. It is not known whether chloroquine reduces the overall number of relapses, or only delays the first relapse. There are many important questions about the biology of vivax malaria of relevance to treatment that remain unanswered. For example is the number of relapses per infection (i.e. per successful inoculation) predetermined or adaptive? If it is predetermined then suppression of the first relapse (as with chloroquine, mefloquine or piperaquine) will reduce the total number of relapses and this is a clear benefit. If it is adaptive then these drugs will simply delay the relapses and there is less clear benefit. These various uncertainties illustrate the importance of detailed comparative longitudinal evaluations. In order to characterize the biology of vivax malaria, it will be necessary to compare regimens with and without primaquine. Because of the challenges that face primaquine prescription (side effects, toxicity in G6PD deficient patients and duration of treatment), it is not commonly deployed along the Thai Burma border. In effect, we will be comparing usual practice (non primaquine regimens) with the recommended WHO and Thai MOPH practice (use of primaquine for 14 days). The information we will gather is crucial to the understanding of chloroquine and its effect on the vivax parasite. This will lead to future studies and invariably change the way we treat vivax malaria.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children > 6 months
* Weight > 7 kg for children
* Have not had primaquine since last Pv episode
* Participant (or parent/guardian if < 18 years old) is willing and able to give written informed consent
* Microscopic diagnosis of Plasmodium vivax mono-infection
* Ability (in the investigators opinion) and willingness of patient or parent/guardian to comply with all study requirements

Exclusion Criteria

* Allergy to artesunate, chloroquine or primaquine
* Severe malaria
* Patients with microscopic diagnosis of co-infection with Plasmodium falciparum
* Presence of any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study
* Inability to tolerate oral medication
* Pregnancy
* Blood transfusion in the last 3 months
* Antimalarial in last 2 months

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The first recurrence of Plasmodium vivax malaria | Day 28
  The first recurrence of Plasmodium vivax malaria within 28 days

SECONDARY OUTCOMES:
Any recurrence of Plasmodium vivax parasitemia | 1 year
  Any recurrence of Plasmodium vivax parasitemia within the follow up period
Time to first recurrence, median time between episodes of vivax infections and total number of episodes | 1 year
  Time to first recurrence, median time between episodes of vivax infections and total number of episodes in the follow up period
Overall number of days of illness and haematocrit below 30% | 1 year
  Overall number of days of illness and haematocrit below 30% within the follow up period
Chloroquine level | Day 7
  Whole blood chloroquine level at day 7 and any day of recurrence of Plasmodium vivax malaria
Adverse events | 1 year
  Adverse event profiles of artesunate, chloroquine and primaquine

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Thailand

REFERENCES:
- [Derived] Stadler E, Cromer D, Mehra S, Adekunle AI, Flegg JA, Anstey NM, Watson JA, Chu CS, Mueller I, Robinson LJ, Schlub TE, Davenport MP, Khoury DS. Population heterogeneity in Plasmodium vivax relapse risk. PLoS Negl Trop Dis. 2022 Dec 19;16(12):e0010990. doi: 10.1371/journal.pntd.0010990. eCollection 2022 Dec. PMID 36534705
- [Derived] Chu CS, Phyo AP, Lwin KM, Win HH, San T, Aung AA, Raksapraidee R, Carrara VI, Bancone G, Watson J, Moore KA, Wiladphaingern J, Proux S, Sriprawat K, Winterberg M, Cheah PY, Chue AL, Tarning J, Imwong M, Nosten F, White NJ. Comparison of the Cumulative Efficacy and Safety of Chloroquine, Artesunate, and Chloroquine-Primaquine in Plasmodium vivax Malaria. Clin Infect Dis. 2018 Oct 30;67(10):1543-1549. doi: 10.1093/cid/ciy319. PMID 29889239
- [Derived] Pratt B, Zion D, Lwin KM, Cheah PY, Nosten F, Loff B. Closing the translation gap for justice requirements in international research. J Med Ethics. 2012 Sep;38(9):552-8. doi: 10.1136/medethics-2011-100301. Epub 2012 Mar 16. PMID 22427705